CLINICAL TRIAL: NCT02549846
Title: Randomized Controlled Trial of Early Versus Late Statin Therapy in Patients With Ischemic Stroke
Brief Title: AdminiStration of Statin On Acute Ischemic stRoke patienT Trial
Acronym: ASSORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Collaborators: Shionogi (Industry)
Responsible Party: Principal Investigator, Shinichi Yoshimura, Principal Investigator, Hyogo Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMIN000021032
Record Dates: First submitted 2015-08-11; First posted 2015-09-15 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute Group (Active Comparator): Atorvastatin 20 mg or Pitavastain 4 mg or Rosuvastatin 5 mg treatment initiated within 24 hours after admission
  Interventions: Drug: Statin
- Stable Group (Other): Not start or withdraw Atorvastatin 20 mg or Pitavastain 4 mg or Rosuvastatin 5 mg treatment for a weak after admission.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Randomized controlled trial of early versus late statin therapy in patients with ischemic stroke
  Other Names: Atorvastatin, Pitavastain, Rosuvastatin

SUMMARY:
Investigators will study whether immediate statin treatment after the onset of stroke is beneficial on the neurological protection

DETAILED DESCRIPTION:
It is much more important in Japan than Western to improve the prognosis after stroke because the prevalence and mortality rate of stroke in Japan is about 3-4 times as those of acute myocardial infarction. Investigators will study whether immediate statin treatment after the onset of stroke is beneficial on the neurological protection since most of previous studies with statins just showed the preventive effects from onset of primary or recurrent cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* the Informed consent will be acquired by the document.
* Age: 20 years of age or older.
* Gender: unquestioned
* hospitalization, outpatient: hospital
* Patients by MRI at the time of hospital transport, it has been confirmed diagnosed with cerebral infarction
* ingestible in within 24 hours after admission In the study treatment period, patients that can be defined treatment in this clinical study implementation plan

Exclusion Criteria:

* patients with a history of hypersensitivity to the treatment agent of the present study
* Patients acute hepatitis, chronic hepatitis acute exacerbation, liver cirrhosis, it is believed that the liver cancer, liver function jaundice or the like is reduced, or a biliary obstruction
* Patients suspected of being pregnant or pregnant
* Patients in the administration of the cyclosporine or telaprevir
* patients with moderate or severe renal impairment (SCr ≧ 2.5mg / dL or eGFR <30mg / dL)
* Patients who received a diagnosis of acute coronary syndrome within 6 months
* valvular disease, atrial fibrillation, patients with atrial thrombus
* Patients familial hypercholesterolemia
* patient admission NIHSS score is greater than or equal to 3 is more than 20 or before the onset mRS score
* patients with other doctors deemed inappropriate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | 12 weeks from stroke onset
  Scale range from 0 [no symptom] to 6 [dead]

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Yoshimura, Principal Investigator — Hyogo collage of Medicine
Locations (1):
- Hyogo collage of Medicine, Nishinomiya, Hyōgo, Japan

REFERENCES:
- [Derived] Yoshimura S, Uchida K, Daimon T, Takashima R, Kimura K, Morimoto T; ASSORT Trial Investigator. Randomized Controlled Trial of Early Versus Delayed Statin Therapy in Patients With Acute Ischemic Stroke: ASSORT Trial (Administration of Statin on Acute Ischemic Stroke Patient). Stroke. 2017 Nov;48(11):3057-3063. doi: 10.1161/STROKEAHA.117.017623. Epub 2017 Oct 13. PMID 29030478